CLINICAL TRIAL: NCT03341403
Title: Assessment of the Impact of a Dietary Supplement Synbiotic "Probiotical ®/Bactecal®" in Asthma
Brief Title: Effect of a Synbiotic "Probiotical®/Bactecal® " in Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Renaud Louis, Professor, University of Liege
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-248; B707201733638 (Other: clinicaltrials.be)
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Asthma
Keywords: severe asthma; synbiotic; immunomodulation; sputum
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: randomized double blind placebo control study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only Phacobel which provide the pills will have the knowledge of the pills codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic group (Active Comparator): severe asthmatic patients (ACQ> 1.5 and beclomethasone > 200 µg per day) will receive "Probiotical ®/Bactecal®" (3 pills a day, content: Lactobacillus, Bifidobacterium et Streptococcus thermophilus, 18 billion of bacteria per pill) during 3 months.
  Interventions: Dietary Supplement: Probiotical®/Bactecal®
- Placebo group (Placebo Comparator): severe asthmatic patients (ACQ> 1.5 and beclomethasone > 200 µg per day) will receive a placebo (3 pills a day) during 3 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotical®/Bactecal® — "Probiotical/Bactecal®" is composed of: Lactobacillus, Bifidobacterium et Streptococcus thermophilus, 18 billion of bacteria per pill.
  Arms: Synbiotic group
Other: Placebo — pills containing placebo
  Arms: Placebo group

SUMMARY:
It is a randomized double blind placebo control study. One hundred severe asthmatic patients will receive "Probiotical ®/Bactecal®" each day during 3 months and will be evaluated before and 1-3-6 months after in order to assess the impact of the synbiotic on the lung function, the exhaled nitric oxide value, the inflammatory blood and sputum profiles, the bronchial reactivity, the microvascular health and the quality of life and asthma control. The hypothesis is that, as these patients are not optimally controlled, the synbiotic could have an impact by decreasing the inflammation state at local and systemic level and then improve the quality of life and the asthma control. Indeed, synbiotic have been shown to possess beneficial effects on the immune system.

DETAILED DESCRIPTION:
Thirty percent of asthmatic patients are not well controlled even with an optimal treatment. There is then a need for new therapeutics allowing a better asthma control. Synbiotic (association of probiotics and prebiotics) have been shown to have anti-inflammatory properties as well as immunomodulatory activities. Moreover, synbiotic appeared to be very well tolerated and safe.

One hundred severe asthmatic patients (ACQ> 1.5 and beclomethasone > 200 µg per day) will receive "Probiotical ®/Bactecal®" (3 pills a day, content: Lactobacillus, Bifidobacterium et Streptococcus thermophilus, 18 billion of bacteria per pill) or a placebo during 3 months.

They will be evaluated before and 1-3-6 months after the first administration and different tests will be realized:

* lung function tests (spirometry, lung volumes, diffusing capacity)
* exhaled nitric oxide value (FeNo, linked to airway eosinophilia)
* blood tests: leucocyte count, c reactive protein, fibrinogen. Plasma and serum will be kept for inflammatory mediators measurements.
* sputum induction: leucocyte count and mediators measurements using the sputum supernatant and sputum cells.
* bronchial reactivity (bronchial challenge test)
* microvascular health: to assess the glycocalyx state, see: http://glycocheck.com/ for details.
* questionnaires: asthma control test (ACT), asthma control questionnaire (ACQ), asthma quality of life questionnaire (AQLQ ).

ELIGIBILITY:
Inclusion Criteria:

* severe asthma (ACQ >1.5 and treatment = minimum 200 µg beclomethasone) and stable treatment for at least 3 months.

Exclusion Criteria:

* treatment not stable
* exacerbation state
* infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
ACQ improvement | before the administration and 1-3-6 months after the first administration
  improvement of asthma control. Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom and bronchodilator use questions on a 7-point scale (0=no impairment, 6= maximum impairment). The questions are equally weighted and the ACQ score is the mean of the 7 questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). An improvement correspond to a decrease of at least 0.5 compared to the last evaluation.

SECONDARY OUTCOMES:
exhaled nitric oxide value decrease | before the administration and 1-3-6 months after the first administration
  measure in ppb with a chemoluminescence analyser

OTHER OUTCOMES:
blood eosinophil count decrease | before the administration and 1-3-6 months after the first administration
  in absolute value
sputum eosinophil count decrease | before the administration and 1-3-6 months after the first administration
  in absolute value
sputum eosinophil percentage decrease | before the administration and 1-3-6 months after the first administration
  in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Louis, Prof., Principal Investigator — CHU-ULG
Locations (1):
- University Hospital of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Glycocheck website — http://glycocheck.com/
- See also: interreg Euregio Meuse Rhine project — https://www.interregemr.eu/projects/healthyaging-en